CLINICAL TRIAL: NCT01930461
Title: A Dose Ranging Study Investigating the Efficacy and Safety of Sublingual Immunotherapy Tablets of House Dust Mite Allergen Extracts in Adults With House Dust Mite-associated Allergic Asthma
Brief Title: Dose Ranging Study of SLIT Tablets of House Dust Mite Allergen Extracts (HDM) in Adults With HDM-associated Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO72.12
Record Dates: First submitted 2013-08-16; First posted 2013-08-29 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Asthma; House Dust Mite Allergy
MeSH Terms: conditions — Asthma; Dust Mite Allergy | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SLIT (A) (Experimental): SLIT tablets of HDM allergen extracts, 3 different doses (A)
  Interventions: Biological: SLIT tablets of HDM allergen extracts, 3 different doses (A)
- SLIT (B) (Experimental): SLIT tablets of HDM allergen extracts, 3 different doses (B)
  Interventions: Biological: SLIT tablets of HDM allergen extracts, 3 different doses (B)
- SLIT (C) (Experimental): SLIT tablets of HDM allergen extracts, 3 different doses (C)
  Interventions: Biological: SLIT tablets of HDM allergen extracts, 3 different doses (C)
- Placebo (Placebo Comparator): Placebo matching the SLIT tablets of HDM allergen extracts
  Interventions: Biological: Placebo matching the SLIT tablets of HDM allergen extracts

INTERVENTIONS:
Biological: SLIT tablets of HDM allergen extracts, 3 different doses (A) — Two sublingual tablets daily for 13 months
  Other Names: Sublingual immunotherapy tablet
  Arms: SLIT (A)
Biological: SLIT tablets of HDM allergen extracts, 3 different doses (B) — Two sublingual tablets daily for 13 months
  Other Names: Sublingual immunotherapy tablet
  Arms: SLIT (B)
Biological: SLIT tablets of HDM allergen extracts, 3 different doses (C) — Two sublingual tablets daily for 13 months
  Other Names: Sublingual immunotherapy tablet
  Arms: SLIT (C)
Biological: Placebo matching the SLIT tablets of HDM allergen extracts — Two sublingual tablets daily for 13 months
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of different doses of sublingual tablets of house dust mite allergen extracts as compared to placebo in adults with house dust mite-associated allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female from 18 to 50 years of age.
* Diagnosed asthma and rhinitis with medical history consistent with HDM-induced allergic asthma and rhinitis.
* Positive SPT to HDM and and HDM-specific IgE serum value ≥ 0.7 kU/L.
* Stable asthma therapies.
* Spirometry (pre-bronchodilator) with best FEV1 ≥ 70% of the predicted value.
* Spirometry with reversibility in FEV1 of ≥ 12% and ≥ 200 mL.
* Asthma Control Test™ (ACT) score ≤ 19.

Exclusion Criteria:

* Former smoker with > 10 pack year history or current smoker.
* Patient with a urine level of cotinine ≥ 500 ng/mL.
* Co-sensitisation to any allergen possibly leading to clinically relevant symptoms likely to significantly change the asthma symptoms of the subject during the study.
* Patient who received allergen immunotherapy for HDM within the past 10 years.
* Ongoing immunotherapy for an aeroallergen other than house dust mite.
* Patient with any oral condition that could confound the safety assessments or planning to have a dental extraction during the study.
* Patient treated with beta-blockers, tricyclic antidepressants or monoamine oxidase inhibitors (MAOIs).
* Pregnant women or breast-feeding/lactating.
* Women with childbearing potential who are not using a medically accepted birth control method.
* Patient with a past or current disease, which as judged by the Investigator, may affect the patient's participation in, or the outcome of this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 386 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Effect on the Asthma control test (ACT) score | 13 months
  Assessment of the effect of one year of treatment of 3 different doses of sublingual immunotherapy tablets of house dust mite (HDM) allergen extracts as compared to placebo on the Asthma Control Test™ (ACT) score, in adults with HDM-associated allergic asthma

SECONDARY OUTCOMES:
Number and percentage of subjects with treatment-emergent AEs | Measured during 13 months

OTHER OUTCOMES:
Changes of Immunological parameters (HDM-specific IgE and IgG4 values) | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Demoly, MD, Principal Investigator — Montpellier, France
Locations (5):
- France (2):
  - CHU Arnaud de Villeneuve, Montpellier
  - NHC, Hôpitaux Universitaires de Strasbourg, Strasbourg
- Universitätsmedizin Berlin - Allergie-Centrum-Charité, Berlin, Germany
- Poland (2):
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 1im.N.Barlickiego w Uniwersystetu Medycznego w Łodzi, Lodz
  - Majorek-Olechowska Bernadetta, Tarnów